CLINICAL TRIAL: NCT03255629
Title: Closed-Loop Glucagon Pump for Treatment of Post-Bariatric Hypoglycemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Xeris Pharmaceuticals (Industry); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-27; 1R44DK107114 (NIH)
Record Dates: First submitted 2017-08-10; First posted 2017-08-21 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Post-bariatric Hypoglycemia
MeSH Terms: interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: A randomization scheme will be devised to assign half the subjects to receive glucagon during their first challenge visit and the other half to receive vehicle during their first challenge visit. At their second challenge subjects will be assigned to the product not received during their first challenge. The label will include a subject randomization number and information as to which vial should be administered during the first challenge and which should be administered during the second challenge.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medication will be provided in vials which are labeled with randomization information only but not contents of vial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Study drug (glucagon) first, placebo second (Other): Each subject will have two mixed meal tolerance tests performed. Each will be randomized to receive either glucagon or matched placebo during the first testing session. A participant could receive 2 doses of the study drug or placebo at each study visit. The opposite treatment will be given during the second testing session after a 1-2 week washout period. Both participants and the study team will be blinded to the intervention being used during each session.
  Interventions: Drug: glucagon; Device: Closed loop glucagon pump
- Placebo first, study drug (glucagon) second (Other): Each subject will have two mixed meal tolerance tests performed. Each will be randomized to receive either glucagon or matched placebo during the first testing session. A participant could receive 2 doses of the study drug or placebo at each study visit. The opposite treatment will be given during the second testing session after a 1-2 week washout period. Both participants and the study team will be blinded to the intervention being used during each session.
  Interventions: Device: Closed loop glucagon pump

INTERVENTIONS:
Drug: glucagon — novel, stable non-aqueous glucagon formulation provided by Xeris Pharmaceuticals
  Arms: Study drug (glucagon) first, placebo second
Device: Closed loop glucagon pump — a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.

SUMMARY:
To assess the efficacy of a closed loop glucagon system to prevent and treat hypoglycemia occurring in patients with Post-Bariatric Hypoglycemia (PBH) in response to meals and exercise.

DETAILED DESCRIPTION:
A control system for sensor-guided delivery was previously developed and tested in a Proof-of-Concept (POC) study in a clinical research setting during 9 mixed meal tolerance tests in 8 unique patients with severe hypoglycemia following bariatric surgery. This optimized algorithm will now be implemented to deliver stable glucagon in a closed-loop system.

A randomized, placebo-controlled, masked trial will be conducted to assess the efficacy of the closed loop system to prevent and treat hypoglycemia occurring in patients with PBH in response to meals (part 1). Part 2 will test whether the closed loop system can also prevent and treat hypoglycemia in patients with PBH in response to exercise. A manufacturing program from our collaborating team at Xeris Pharmaceuticals will continue to produce supplies of glucagon for the clinical trial in a current good manufacturing practice (cGMP) facility, with continued shelf-life stability testing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females diagnosed with ongoing post-bariatric hypoglycemia with prior episodes of neuroglycopenia, unresponsive to dietary intervention (low glycemic index, controlled carbohydrate portions) and trial of acarbose therapy at the maximally tolerated dose.
2. Age 18-65 years of age, inclusive, at screening.
3. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion Criteria:

1. Documented hypoglycemia occurring in the fasting state (> 12 hours fast);
2. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
3. Hepatic disease, including serum alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
4. Congestive heart failure, New York Heart Association (NYHA )class II, III or IV;
5. History of myocardial infarction, unstable angina or revascularization within the past 6 months or 2 or more risk factors for coronary artery disease including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use;
6. History of cardiac arrhythmia or arrhythmia detected by EKG during the screening visit;
7. History of syncope (unrelated to hypoglycemia) or diagnosed cardiac arrhythmia
8. Concurrent administration of β-blocker therapy;
9. History of a cerebrovascular accident;
10. Seizure disorder (other than with suspect or documented hypoglycemia);
11. Active treatment with any diabetes medications except for acarbose;
12. Active malignancy, except basal cell or squamous cell skin cancers;
13. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma (MEN 2, neurofibromatosis, or Von Hippel-Lindau disease);
14. Known insulinoma or glucagonoma;
15. Major surgical operation within 30 days prior to screening;
16. Hematocrit < 33%;
17. Bleeding disorder, treatment with warfarin, or platelet count <50,000;
18. Blood donation (1 pint of whole blood) within the past 2 months;
19. Active alcohol abuse or substance abuse;
20. Current administration of oral or parenteral corticosteroids;
21. Pregnancy and/ or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intrauterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence;
22. Use of an investigational drug within 30 days prior to screening;
23. Current use of anticholinergic medications;
24. Allergy to a component of the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulla CM, Zavitsanou S, Laguna Sanz AJ, Pober D, Richardson L, Walcott P, Arora I, Newswanger B, Cummins MJ, Prestrelski SJ, Doyle FJ, Dassau E, Patti ME. A Randomized, Placebo-Controlled Double-Blind Trial of a Closed-Loop Glucagon System for Postbariatric Hypoglycemia. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1260-71. doi: 10.1210/clinem/dgz197. PMID 31714583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a history of Roux-en-Y gastric bypass (RYGB) and post-bariatric hypoglycemia (PBH) with neuroglycopenia, uncontrolled on medical nutrition therapy and medications, were recruited from the Joslin Diabetes Center hypoglycemia clinic and other endocrine clinics in the region.
Pre-assignment Details: Between September 2017 and August 2018, 23 individuals were screened and 18 enrolled (consort diagram, Fig. 2). Two participants withdrew before the first mixed-meal study visit because of inability to obtain adequate intravenous access.
Groups:
- Study Drug (Glucagon) First, Then Placebo (Randomized, Double-blind, Crossover Design): Each subject underwent two mixed meal tolerance tests, and was randomized to receive either glucagon or placebo during the first testing session (opposite treatment was given during the second testing session). These participants received glucagon first, and then the placebo at the second visit. A participant could receive 2 doses of the study drug or placebo at each study visit.
  Glucagon: novel, stable, non-aqueous glucagon formulation provided by Xeris Pharmaceuticals.
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
- Placebo First, Then Study Drug (Glucagon) Second (Randomized, Double-blind, Crossover Design): Each subject underwent two mixed meal tolerance tests performed. Each was randomized to receive either glucagon or matched placebo during the first testing session. The opposite treatment was given during the second testing session. Both participants and the study team were blinded to the intervention being used during each session.
  These participants received placebo at the fist visit, and the study drug glucagon at the second visit. A participant could receive 2 doses of the study drug or placebo at each study visit.
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation (for this group - they received placebo first) together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
Period: Overall Study
Arm/Group | Study Drug (Glucagon) First, Then Placebo (Randomized, Double-blind, Crossover Design) | Placebo First, Then Study Drug (Glucagon) Second (Randomized, Double-blind, Crossover Design)
Started | 8 | 8
Completed | 5 (One participant developed intractable nausea and emesis after consuming the mixed meal, and was withdrawn. Two participants were withdrawn due to not experiencing hypoglycemia during mixed meal testing.) | 7 (One participant was withdrawn due to not experiencing hypoglycemia during mixed meal testing.)
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — did not experience hypoglycemia | 2 | 1

BASELINE CHARACTERISTICS:
Population: Demographic Information for 12 Enrolled Participants Who Completed 2 Mixed-Meal Study Visits and Were Included in the Analysis
Groups:
- Treatment Arm / Control Arm (Randomized, Double-Blind, Placebo-Controlled Crossover Design): Each subject will have two mixed meal tolerance tests performed. Each will be randomized to receive either glucagon or matched placebo during the first testing session. The opposite treatment will be given during the second testing session. Both participants and the study team will be blinded to the intervention being used during each session.
  glucagon: novel, stable non-aqueous glucagon formulation provided by Xeris Pharmaceuticals
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
Arm/Group | Treatment Arm / Control Arm (Randomized, Double-Blind, Placebo-Controlled Crossover Design)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (1.5)
Years since surgery [Mean (Standard Deviation); unit: years] | 8.4 (1.5)
Years from surgery to neuroglycopenia [Median (Inter-Quartile Range); unit: years] | 2.2 [1.4 to 6.1]
HbA1c [Mean (Standard Deviation); unit: percent] | 5.3 (0.1)
On any anti-hypoglycemic medications [Count of Participants; unit: Participants] | 10
Treated with acarbose [Count of Participants; unit: Participants] | 5
Treated with diazoxide [Count of Participants; unit: Participants] | 4
Treated with octreotide [Count of Participants; unit: Participants] | 3
Treated with pramlintide [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Meal-provoked Hypoglycemia, Defined as Sensor Glucose <65 mg/dL
Description: A primary endpoint for this study is the prevention of meal provoked hypoglycemia, defined as sensor glucose levels below <65 mg/dl, comparing study drug to control.
Time Frame: Measured following 2 challenges: 1 with glucagon and 1 with vehicle. The second challenge was conducted within two weeks of the first.
Population: 12 Enrolled Participants Completed 2 Mixed-Meal Study Visits and Were Included in the Analysis
Measure: Number; unit: participants
Groups:
- Study Drug (Glucagon) Phase: This phase represents when the participant received the study drug - glucagon. A participant could receive 2 doses of the study drug at this visit.
  Each subject had two mixed meal tolerance tests performed. Each was randomized to receive either glucagon or matched placebo during the first testing session. The opposite treatment was given during the second testing session after a 1-2 wk washout period. Both participants and the study team were blinded to the intervention being used during each session.
  glucagon: novel, stable non-aqueous glucagon formulation provided by Xeris Pharmaceuticals
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
- Placebo / Control Phase: This phase represents when the participant received the placebo. A participant could receive 2 doses of the placebo at this visit.
  Each subject had two mixed meal tolerance tests performed. Each was randomized to receive either glucagon or matched placebo during the first testing session. The opposite treatment was given during the second testing session after a 1-2 week washout period. Both participants and the study team were blinded to the intervention being used during each session.
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation (for this phase containing placebo vs. glucagon) together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
participants | 1 | 5
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.103, McNemar

2. Primary Outcome: Number of Participants With Meal-provoked Hypoglycemia, Defined as Plasma Glucose <65 mg/dL
Description: A primary endpoint for this study is prevention of meal provoked hypoglycemia, defined as plasma glucose levels below <65 mg/dl, comparing study drug to control
Time Frame: as for outcome 1
Population: Measured following 2 challenges: 1 with glucagon and 1 with vehicle. The second challenge was conducted within two weeks of the first.
Measure: Count of Participants; unit: Participants
Groups:
- Study Drug (Glucagon) Phase: This phase represents when the participant received the study drug - glucagon. A participant could receive 2 doses of the study drug at this visit.
  Each subject had two mixed meal tolerance tests performed. Each was randomized to receive either glucagon or matched placebo during the first testing session. The opposite treatment was given during the second testing session after a 1-2 week washout period. Both participants and the study team were blinded to the intervention being used during each session.
  glucagon: novel, stable non-aqueous glucagon formulation provided by Xeris Pharmaceuticals
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
Participants | 1 | 4
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.180, McNemar

3. Secondary Outcome: Number of Participants With Meal-provoked Hypoglycemia, Defined as Sensor Glucose <60 mg/dL
Description: Prevention of meal / provoked hypoglycemia, defined as sensor glucose levels below <60 mg/dl, comparing vehicle to control
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
Participants | 1 | 3

4. Secondary Outcome: Number of Participants With Rebound Hyperglycemia (Defined as Glucose Levels Above 180 mg/dl).
Description: Compare outcomes for glucagon versus vehicle infusions for prevention of rebound hyperglycemia (defined as glucose levels above 180 mg/dl).
Time Frame: Measured following 2 challenges: 1 with glucagon and 1 with vehicle. The second challenge will be conducted within two weeks of the first.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.317, McNemar

5. Secondary Outcome: Number of Participants With Hypoglycemia Rescue Administered
Description: Protocol-specified rescue delivery of IV glucose was performed if plasma glucose <55 mg/dL and/or significant neuroglycopenia developed.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
Participants | 0 | 7
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.008, McNemar

6. Secondary Outcome: Number of Participants With Meal-provoked Hypoglycemia, Defined as Plasma Glucose <60 mg/dL
Description: Prevention of meal / provoked hypoglycemia, defined as plasma glucose levels below <60 mg/dl, comparing vehicle to control
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
Participants | 0 | 3
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.083, McNemar

7. Secondary Outcome: Number of Participants With Meal-provoked Hypoglycemia, Defined as Plasma Glucose <55 mg/dL
Description: Prevention of meal / provoked hypoglycemia, defined as plasma glucose levels below <55 mg/dl, comparing vehicle to control
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
Participants | 0 | 5
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.025, McNemar

8. Secondary Outcome: Number of Participants With Meal-provoked Hypoglycemia, Defined as Sensor Glucose <55 mg/dL
Description: Prevention of meal / provoked hypoglycemia, defined as sensor glucose levels below <55 mg/dl, comparing vehicle to control
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

9. Secondary Outcome: Percent Time Plasma Glucose in Range After the Final Dose of Study Drug or Vehicle, Which Was Either 1 or 2 Doses Depending on Patient Response
Description: Compare outcomes for glucagon versus vehicle infusions for percent time plasma glucose in range (180-65mg/dL) after the final dose, which was either 1 or 2 doses depending on patient response
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
percentage of time | 0.852 (0.082) | 0.645 (0.074)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.049, Mixed Models Analysis; Linear mixed effects models to account for correlation within subjects over time

10. Secondary Outcome: Percent Time Sensor Glucose in Range After Drug Delivery After the Final Dose of Study Drug or Vehicle, Which Was Either 1 or 2 Doses Depending on Patient Response
Description: Compare outcomes for glucagon versus vehicle infusions for percent time sensor glucose in range (180-65mg/dL) after the final dose, which was either 1 or 2 doses depending on patient response
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
percentage of time | 0.987 (0.013) | 0.815 (0.077)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.056, Mixed Models Analysis; Linear mixed effects models to account for correlation within subjects over time

11. Secondary Outcome: Meal Provoked Nadir Plasma Glucose
Description: Nadir plasma glucose (mg/dl) during meal testing, comparing vehicle to control
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 67.4 (2.70) | 58.5 (1.87)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.004, Mixed Models Analysis

12. Secondary Outcome: Meal Provoked Nadir Sensor Glucose
Description: Nadir sensor glucose (mg/dl) during meal testing, comparing vehicle to control
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 72.7 (2.21) | 65.3 (1.85)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.059, Mixed Models Analysis

13. Secondary Outcome: Time to Nadir Plasma Glucose After Mixed Meal (Min)
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
minutes | 138 (11.9) | 125 (7.43)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.195, Mixed Models Analysis

14. Secondary Outcome: Time to Nadir Sensor Glucose After Mixed Meal (Min)
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
minutes | 156 (11.6) | 134 (6.04)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.043, Mixed Models Analysis

15. Secondary Outcome: Time to Alarm During Mixed Meal Testing (Minutes)
Description: Time to alarm represents the time for the first alarm to occur during mixed meal testing. Alarms are triggered by hypoglycemia (sensor glucose < 65 mg/dL), or by the algorithm predicting that hypoglycemia will occur in less than 30 minutes (taking into account current sensor glucose level (between 65-150 mg/dL) and the rate of change of a rapidly falling sensor glucose level). In the latter case, the alarm is activated even if glucose levels are within the normoglycemic range to allow early detection and response. During both glucagon and vehicle treatment visits, all participants received either 300 μg of glucagon or the equivalent volume of vehicle with the first alarm.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Groups:
- Placebo / Control Arm: This phase represents when the participant received the placebo. A participant could receive 2 doses of the placebo at this visit.
  Each subject had two mixed meal tolerance tests performed. Each was randomized to receive either glucagon or matched placebo during the first testing session. The opposite treatment was given during the second testing session after a 1-2 week washout period. Both participants and the study team were blinded to the intervention being used during each session.
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation (for this phase containing placebo vs. glucagon) together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Arm
Number analyzed (Participants) | 12 | 12
minutes | 89.9 (3.90) | 87.7 (4.9975)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Arm; Test type: Other; p = 0.659, Mixed Models Analysis

16. Secondary Outcome: Time to Delivery (Min)
Description: Time to delivery (min) of study drug during mixed meal testing
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
minutes | 94 (5.52) | 89.3 (5.33)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.406, Mixed Models Analysis

17. Secondary Outcome: Sensor Glucose at Time of Alarm 1 During Mixed Meal Testing (mg/dL)
Description: This is the sensor glucose at which time the first alarm occurred during the mixed meal testing. Alarms are triggered by hypoglycemia (sensor glucose < 65 mg/dL), or by the algorithm predicting that hypoglycemia will occur in less than 30 minutes (taking into account current sensor glucose level (between 65-150 mg/dL) and the rate of change of a rapidly falling sensor glucose level). In the latter case, the alarm is activated even if glucose levels are within the normoglycemic range to allow early detection and response. During both glucagon and vehicle treatment visits, all participants received either 300 μg of glucagon or the equivalent volume of vehicle with the first alarm.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 134 (5.93) | 139 (4.92)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.611, Mixed Models Analysis

18. Secondary Outcome: Capillary Glucose at Time of Alarm 1 During Mixed Meal Testing (mg/dL)
Description: This is the capillary glucose at which time the first alarm occurred during the mixed meal testing. Alarms are triggered by hypoglycemia (sensor glucose < 65 mg/dL), or by the algorithm predicting that hypoglycemia will occur in less than 30 minutes (taking into account current sensor glucose level (between 65-150 mg/dL) and the rate of change of a rapidly falling sensor glucose level). In the latter case, the alarm is activated even if glucose levels are within the normoglycemic range to allow early detection and response. During both glucagon and vehicle treatment visits, all participants received either 300 μg of glucagon or the equivalent volume of vehicle with the first alarm.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 98.1 (7.30) | 109 (5.75)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.183, Mixed Models Analysis

19. Secondary Outcome: Sensor Glucose at Time of Alarm 2 During Mixed Meal Testing (mg/dL)
Description: This is the sensor glucose at which time the second alarm occurred during the mixed meal testing. Alarms are triggered by hypoglycemia (sensor glucose < 65 mg/dL), or by the algorithm predicting that hypoglycemia will occur in less than 30 minutes (taking into account current sensor glucose level (between 65-150 mg/dL) and the rate of change of a rapidly falling sensor glucose level). In the latter case, the alarm is activated even if glucose levels are within the normoglycemic range to allow early detection and response. During both glucagon and vehicle treatment visits, all participants received either 300 μg of glucagon or the equivalent volume of vehicle with the first alarm.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Arm
Number analyzed (Participants) | 12 | 12
mg/dL | 85.7 (4.96) | 70.1 (2.26)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Arm; Test type: Other; p = 0.009, Mixed Models Analysis

20. Secondary Outcome: Capillary Glucose at Time of Alarm 2 During Mixed Meal Testing (mg/dL)
Description: This is the capillary glucose at which time the second alarm occurred during the mixed meal testing. Alarms are triggered by hypoglycemia (sensor glucose < 65 mg/dL), or by the algorithm predicting that hypoglycemia will occur in less than 30 minutes (taking into account current sensor glucose level (between 65-150 mg/dL) and the rate of change of a rapidly falling sensor glucose level). In the latter case, the alarm is activated even if glucose levels are within the normoglycemic range to allow early detection and response. During both glucagon and vehicle treatment visits, all participants received either 300 μg of glucagon or the equivalent volume of vehicle with the first alarm.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
mg/dL | 94.2 (1.70) | 91.7 (8.62)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.789, Mixed Models Analysis

21. Secondary Outcome: Pain Score at Time of First Dose Delivery of Study Drug, Versus Pain Score at Time of First Dose Delivery of Placebo (Comparing First Delivery Pain Scores for Visit Where Participant Received Study Drug vs. Visit Where Participant Received Placebo).
Description: Pain score was assessed verbally, 1 is the least pain (none), 10 is the most severe pain. Pain score at the time of the first administration was compared for the visit where the participant received the study drug vs. the visit where the participant received the placebo. A participant could receive 2 doses of the study drug or placebo at each visit. All 12 participants completed both the study drug phase and the placebo phase. The pain scores for the first administration of study drug vs. first administration of placebo for these two visits were compared. Whether the participant was assigned to the study drug glucagon (vs. placebo) at the first or second MMTT was determined by randomization.
Time Frame: The two study visits where participants were administered either study drug or placebo took place over 2 weeks (there was a 1 to 2 week washout period between visits).
Measure: Mean (Standard Error); unit: pain score
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
pain score | 4.00 (0.685) | 3.83 (0.815)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.865, McNemar

22. Secondary Outcome: Pain Score at Time of Second Dose Delivery of Study Drug, Versus Pain Score at Time of Second Dose Delivery of Placebo (Comparing Second Delivery Pain Scores for Visit Where Participant Received Study Drug vs. Visit Where Participant Received Placebo).
Description: Pain score was assessed verbally, 1 is the least pain (none), 10 is the most severe pain. Pain score at the time of the second administration was compared for the visit where the participant received the study drug vs. the visit where the participant received the placebo. A participant could receive 2 doses of the study drug or placebo at each visit. All 12 participants completed both the study drug phase and the placebo phase. The pain scores from the second administration of study drug vs. second administration of placebo for these two visits were compared. Whether the participant was assigned to the study drug glucagon (vs. placebo) at the first or second MMTT was determined by randomization.
Time Frame: as for outcome 21
Measure: Mean (Standard Error); unit: pain score
Arm/Group | Study Drug (Glucagon) Phase | Placebo / Control Phase
Number analyzed (Participants) | 12 | 12
pain score | 1.14 (0.615) | 1.31 (0.671)
Statistical Analysis 1: Comparison: Study Drug (Glucagon) Phase vs Placebo / Control Phase; Test type: Other; p = 0.875, McNemar

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the the duration of each individuals participation, a 2 to 3 week period of time, encompassing the time of enrollment, to the completion of visit 5.
Description: Regarding discrepancy between participant flow and number of participants at risk: 18 participants enrolled, however two participants withdrew before the first mixed-meal study visit because of inability to obtain adequate intravenous access. Sixteen participants completed the first mixed-meal study visit; 12 participants completed both mixed meal study visits and were included in analysis.
Groups:
- Treatment Arm and Control Arm (Randomized, Double-Blind, Placebo-Controlled Crossover Design): Each subject had two mixed meal tolerance tests performed. Each was randomized to receive either glucagon or matched placebo during the first testing session. The opposite treatment was given during the second testing session. Both participants and the study team were blinded to the intervention being used during each session.
  glucagon: novel, stable non-aqueous glucagon formulation provided by Xeris Pharmaceuticals
  Closed loop glucagon pump: a novel closed-loop glucagon system (CLG) incorporating a novel, stable non-aqueous glucagon formulation together with an infusion pump system (Omnipod) guided by real-time continuous glucose monitoring (Dexcom) that is triggered by a hypoglycemia alert algorithm.
Arm/Group | Treatment Arm and Control Arm (Randomized, Double-Blind, Placebo-Controlled Crossover Design)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm and Control Arm (Randomized, Double-Blind, Placebo-Controlled Crossover Design) (N=18)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) — Pt was not randomized. hypokalemia discovered during screening visit; admitted to hospital. resolved without sequelae. not related to study protocol or intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm and Control Arm (Randomized, Double-Blind, Placebo-Controlled Crossover Design) (N=18)
Hyperkalemia at screening visit (Metabolism and nutrition disorders) | 1 (1) — Discovered at screening visit. No treatment. Labs were repeated at Visit 2, potassium was within reference range.
MCH above normal limit of refrence range at screening visit. (Blood and lymphatic system disorders) | 1 (1) — No treatment. Complete blood count (CBC) repeated on 2/28/2018.Labs were acceptable to begin study visit.
WBC above normal limit of reference range at screening visit (Blood and lymphatic system disorders) | 1 (1) — No treatment. CBC repeated on 2/28/2018.Labs were acceptable to begin study visit.
Headache prior to start of MMTT (General disorders) | 2 (2) — Not related to study drug or placebo as was present upon arrival.
Tiredness prior to start of MMTT (General disorders) | 1 (1) — Not related to study drug or placebo as was present upon arrival to study visit.
Nausea after intake of mixed meal (prior to glucagon OR placebo) (Gastrointestinal disorders) | 12 (16) — Related to mixed meal tolerance test (MMTT). Resolved without sequelae.
Headache after intake of mixed meal (prior to glucagon OR placebo) (General disorders) | 7 — Related to MMTT. Resolved without sequelae.
Palpitations after intake of mixed meal (prior to study drug OR placebo) (Cardiac disorders) | 6 — Related to MMTT. Resolved without sequelae.
Emesis after intake of mixed meal (prior to study drug OR placebo) (Gastrointestinal disorders) | 2 — Adverse event (AE) linked to meal tolerance test, especially in patient population under study. Required ER evaluation in 1 participant due to repetitive vomiting. All resolved.
Feeling cold / chills after intake of mixed meal (prior to study drug OR placebo) (General disorders) | 3 — Related to MMTT, resolved.
Feeling hot / warm after intake of mixed meal (prior to study drug or placebo) (General disorders) | 6 — AE linked to MMTT. Resolved.
Thirsty after intake of mixed meal (prior to study drug OR placebo) (General disorders) | 1 (1) — Related to MMTT. Resolved.
Tiredness after intake of mixed meal (prior to study drug OR placebo) (General disorders) | 11 — AE linked to MMTT. Resolved.
Stomach ache / cramping after intake of mixed meal (prior to study drug OR placebo) (Gastrointestinal disorders) | 2 — AE linked to MMTT. Resolved.
Bloated / uncomfortably full after intake of mixed meal (prior to study drug OR placebo) (Gastrointestinal disorders) | 1 (2) — AE linked to MMTT. Resolved.
Blurry vision after intake of mixed meal (prior to study drug OR placebo) (Eye disorders) | 1 — AE linked to MMTT. Resolved.
Tingling (paresthesia) in shoulders after intake of mixed meal (prior to study drug or placebo) (General disorders) | 1 — Related to MMTT. Resolved.
Tingling (paresthesia) around the mouth after intake of mixed meal (prior to study drug or placebo) (General disorders) | 1 — AE linked to MMTT. Resolved.
Dizzy after intake of mixed meal (prior to study drug OR placebo) (General disorders) | 1 — AE linked to MMTT. Resolved.
Feeling unwell ("icky... drunk") after intake of mixed meal (prior to study drug OR placebo) (General disorders) | 1 — AE linked MMTT. Resolved.
Tearful after intake of mixed meal (prior to study drug OR placebo) (General disorders) | 1 — AE linked to MMTT. Resolved.
Pain at pump site during MMTT (prior to delivery of study drug or placebo) (General disorders) | 2 — Related to study device. Resolved.
Pruritis at pump insertion site during MMTT (prior to delivery of study drug or placebo) (Skin and subcutaneous tissue disorders) | 2
Irritation / pain at IV site with IV administration of dextrose (General disorders) | 1 — AE related to administration of D50 at placebo visit. Resolved.
Tearful when IV dextrose (D50) administered (General disorders) | 1 — Related to MMTT & hypoglycemia, at visit where placebo was administered. Resolved.
Hypoglycemia during study (MMTT) (Endocrine disorders) | 13 (21) — Related to MMTT in population understudy. Resolved.
Erythema at site of CGM sensor (Skin and subcutaneous tissue disorders) | 1 — Related to continuous glucose monitoring (CGM) device (sensor or adhesive). Resolved.
Hematoma under CGM sensor (Skin and subcutaneous tissue disorders) | 1 — AE related to CGM sensor device.
Burning pain / pricking at pump site after alarm (placebo visit) (General disorders) | 10 — AE linked to placebo and study device.
Buring pain at pump site after alarm (glucagon visit) (General disorders) | 13
Erythema at pump infusion site (placebo visit) (Skin and subcutaneous tissue disorders) | 10 — AE related to study device and placebo.
Erythema at pump infusion site (glucagon visit) (Skin and subcutaneous tissue disorders) | 11 — AE related to study device and study drug - glucagon.
Edema at pump infusion site (placebo visit) (Skin and subcutaneous tissue disorders) | 4 — AE related to study device and placebo.
Edema at pump infusion site (glucagon visit) (Skin and subcutaneous tissue disorders) | 6 — AE related to study device and study drug - glucagon.
Feeling hot after alarm (glucagon visit) (General disorders) | 2 — AE linked to MMTT, hypoglycemia, and delivery of study drug.
Feeling hot after alarm (placebo visit) (General disorders) | 3 — AE linked to MMTT, hypoglycemia, and delivery of placebo.
Thirsty after alarm (placebo visit) (Endocrine disorders) | 1 — AE linked to MMTT, hypoglycemia, and delivery of placebo.
Nausea after alarm (glucagon visit) (Gastrointestinal disorders) | 1 — AE linked to MMTT, hypoglycemia, and delivery of study drug.
Vomiting after alarm (glucagon visit) (Gastrointestinal disorders) | 1 — Participant also vomited during mixed meal, prior to study drug administration. AE linked to MMTT, hypoglycemia, and delivery of study drug.
Headace after alarm (glucagon visit) (General disorders) | 2 — Both participants with headache following alarm also had headache prior to the alarm during mixed meal testing. AE related to MMTT, hypoglycemia, and study drug - glucagon.
Tearful during alarm (placebo visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Confusion after alarm (placebo visit) (Nervous system disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Confusion after alarm (glucagon visit) (Nervous system disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Dizzy / lightheaded after alarm (glucagon visit) (General disorders) | 2 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Low blood pressure after alarm (placebo visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Tiredness after alarm (glucagon visit) (General disorders) | 2 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Tiredness after alarm (placebo visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Blurry vision after alarm (placebo visit) (Eye disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Blurry vision after alarm (glucagon visit) (Eye disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Bowel urgency after alarm (glucagon visit) (Gastrointestinal disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Bowel movement after alarm (placebo visit) (Gastrointestinal disorders) | 1 — AE related to MMTT, and placebo.
Stomach cramping / pain after alarm (placebo visit) (Gastrointestinal disorders) | 2 — AE related to MMTT and placebo.
Lower extremity cramping after alarm (glucagon visit) (Musculoskeletal and connective tissue disorders) | 2 — Legs and toes cramping. AE related to MMTT, hypoglycemia, and study drug - glucagon.
Pale after alarm (placebo visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Speech slowed after alarm (placebo visit) (Nervous system disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Nausea prior to lunch (glucagon visit) (Gastrointestinal disorders) | 1 — This participant was also nauseous after intake of mixed meal, prior to receiving the study drug. AE related to MMTT, hypoglycemia, and study drug - glucagon.
Weakness prior to lunch (glucagon visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Feeling hot prior to lunch (glucagon visit) (General disorders) | 1 — This participant also felt hot following intake of mixed meal, prior to delivery of study drug. AE related to MMTT, hypoglycemia, and study drug - glucagon.
Feeling hot after lunch (placebo visit) (General disorders) | 2 — AE related to MMTT, hypoglycemia, placebo.
Tiredness after lunch (glucagon visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Tiredness after lunch (placebo visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Feeling cold after lunch (glucagon visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Headache after lunch (glucagon visit) (General disorders) | 2 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Stomach pains after lunch (glucagon visit) (Gastrointestinal disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Nausea after lunch (glucagon visit) (Gastrointestinal disorders) | 1 — Participant also had nausea after intake of mixed meal, prior to delivery of study drug. AE related to MMTT, hypoglycemia, and study drug - glucagon.
Vomiting after lunch (glucagon visit) (Gastrointestinal disorders) | 1 — This participant had nausea which started after intake of mixed meal, prior to study drug administration. AE related to MMTT, hypoglycemia, and study drug - glucagon.
Shaky following lunch (glucagon visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Ears ringing after lunch (General disorders) | 1 — AE related to MMTT. Resolved.
Foggy feeling after lunch (glucagon visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Hypoglycemia following lunch (gluagon visit) (Endocrine disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Hypoglycemia following lunch (placebo visit) (Endocrine disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Back pain after lunch (placebo visit) (Musculoskeletal and connective tissue disorders) | 1 — Not related. Participant with chronic back pain.
Dry mouth following alarm (glucagon visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Pruritis at pump site after alarm (placebo visit) (Skin and subcutaneous tissue disorders) | 1 — AE related to study device and placebo.
Dizzy after discharge (placebo visit) (General disorders) | 1 — AE related to MMTT, hypoglycemia, and placebo.
Hypoglycemia after dinner the night following the study visit (glucagon visit) (Endocrine disorders) | 1 — Possibly related to study visit and study drug (glucagon).
Tiredness day after study visit (placebo visit) (Gastrointestinal disorders) | 3 — AE related to MMTT, hypoglycemia, and placebo.
Tiredness day after study visit (glucagon visit) (General disorders) | 4 — AE related to MMTT, hypoglycemia, and study drug - glucagon.
Migraine headache one night following study visit (placebo visit) (Nervous system disorders) | 1 — Possibly related to MMTT, hypoglycemia, and placebo.
Erythema a pump infusion site 1 day following discharge (glucagon visit) (Skin and subcutaneous tissue disorders) | 1 — 2" diameter corresponding with area of the adhesive. AE related to pump device adhesive. This participant had erythema as well documented on the day of the study visit. Resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT03255629/Prot_SAP_000.pdf